CLINICAL TRIAL: NCT00924898
Title: CID 0805 - Treatment of Acute HIV Infection With a Once Daily Regimen of Emtricitabine, Tenofovir and Efavirenz - A Pilot Study of Response to Therapy and HIV Pathogenesis
Brief Title: Treatment of Acute HIV With Emtricitabine, Tenofovir and Efavirenz (CID 0805)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Bristol-Myers Squibb (Industry); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Cynthia L Gay, MD, Clinical Assistant Professor, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CID 0805 (PHI 02)
Record Dates: First submitted 2009-06-17; First posted 2009-06-19 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Acute HIV Infection; HIV Infections
Keywords: Acute HIV; HIV; Acute Infections; Acute Infection
MeSH Terms: conditions — HIV Infections | interventions — efavirenz; Emtricitabine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acute HIV Treatment Group (Experimental): Single arm, open label study in which all participants received the same study treatment with efavirenz, emtricitabine, and tenofovir DF
  Interventions: Drug: efavirenz, emtricitabine, and tenofovir

INTERVENTIONS:
Drug: efavirenz, emtricitabine, and tenofovir — Once daily ART with emtricitabine, tenofovir DF and efavirenz
  Other Names: Tenofovir disoproxil fumarate; Emtricitabine; FDC Emtricitabine 200 mg/ tenofovir 300 mg; Efavirenz; FDC Emtricitabine 200mg/Tenofovir 300mg DF/Efavirenz 600mg

SUMMARY:
This is a pilot study of treatment of acute HIV infection with a once daily regimen of Emtricitabine, Tenofovir and Efavirenz. The primary objectives of this study are:

1. To determine the safety and tolerability, and the virologic and immunologic efficacy of FTC, TDF, and efavirenz given once daily to patients with acute HIV infection.
2. To assess the impact of once daily therapy combined with a standardized adherence program on treatment adherence, virologic suppression, and rate of viral load decline in blood and infectious fluids (semen, cervico-vaginal secretions).
3. To define the prevalence of genotypic and phenotypic resistance to antiretroviral agents among persons diagnosed with acute HIV infection in the Southeastern United States.

DETAILED DESCRIPTION:
Hypothesis: Once daily ART with fixed dose combination FTC/TDF/EFV will reduce viral replication to <200 copies RNA/ml plasma in blood and other body compartments in patients with acute HIV infection, reducing infectivity. The treatment regimen will be well tolerated during treatment follow-up. A coordinated program of counseling and support will facilitate adherence and promote successful therapy. Prevalence of transmitted drug resistant HIV-1 will be assessed.

Study Design: Dual-center, prospective, single-arm pilot study of FTC/TDF/EFV in patients with acute HIV infection. Study sites will be members of the Duke-UNC Acute HIV Infection Study Consortium. Patients will be followed intensively for 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of acute HIV infection as defined by protocol.
2. The following laboratory parameters verified within 30 days of study entry:

   * Bilirubin </= 3.0mg/dL
   * ALT/AST </= 10 X upper limit of normal
   * Absolute neutrophil count (ANC) >/= 500cells/mm3
   * Platelet count >/= 25,000 cells/mm3
   * Hemoglobin >/= 8.5g/dL for men and >/= 8.0 g/dL for women
   * Calculated creatinine clearance (Cockcroft-Gault formula) >/= 50mL/min:

   CrCl = (140-age) x body weight (kg) (x 0.85 if female)/ Serum creatinine [mg/dL] x (72)
3. All women of child-bearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of bHCG) within 72 hours prior to start of study medication. WOCBP is defined as any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), who is not postmenopausal (defined as amenorrhea >/=12 consecutive months), or is on hormone replacement therapy (HRT) with documented plasma follicle-stimulating hormone level >/=35mLU/mL. Women who are using oral, implanted, or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child bearing potential;
4. Be willing to use two effective forms of contraception throughout study. Barrier contraception should always be used in combination with other methods of contraception (oral or other hormonal contraceptives);
5. Weigh >/= 40 kg;

Exclusion Criteria:

1. A life expectancy less than twelve months.
2. Women who are pregnant or breastfeeding.
3. Women with a positive pregnancy test on enrollment or prior to study drug administration.
4. WOCBP who are unwilling or unable to use two acceptable methods to avoid pregnancy for the entire study period
5. WOCBP using a prohibited contraceptive method
6. Hypersensitivity to any component of the formulation of study drugs.
7. A clinically important illness not explicitly excluded by the protocol, a physical or psychiatric disability, or a laboratory abnormality that might place the patient at increased risk by being exposed to the medications in this study or which might confound the interpretation of this investigation.
8. Proven or suspected acute hepatitis within 30 days prior to study entry (this excludes liver inflammation related to acute HIV infection).
9. Intractable diarrhea (>/=6 loose stools/day for at least 7 consecutive days) within 30 days prior to study entry or vomiting lasting more than 4 days within one month prior to dosing (this excludes symptoms attributed to acute HIV infection).
10. An active AIDS-defining opportunistic infection or disease (for the purpose of this study, a CD4 count </=200 cells/mm3 in the absence of any other AIDS-defining indicator condition is not considered an AIDS-defining event. AIDS-defining events occurring during the acute HIV infection syndrome period such as Candida esophagitis will be considered on a case-by-case basis and will not be automatically considered exclusionary).
11. Inability to communicate effectively with study personnel.
12. Current alcohol or recreational drug use which in the investigator's opinion interferes with the subject's ability to comply with dosing schedule and protocol evaluations or increases the risk of developing pancreatitis.
13. Incarceration; prisoner recruitment and participation are not permitted.
14. Difficulty swallowing capsules/tablets.
15. Prior treatment with any other experimental drug for any indication (within 30 days of initiating study treatment).
16. Treatment with immune-modulating agents (within 30 days of initiating study treatment) such as cyclosporine and systemic corticosteroids. Routine vaccinations are allowed.
17. Therapy with agents with significant systemic neurotoxic pancreotropic or cytotoxic potential within 3 months of study start, or the need for such therapy is expected at the time of enrollment.
18. Therapy with nephrotoxic agents (aminoglycosides, IV amphotericin, cidofovir, IV pentamidine, cisplatin other agents with nephrotoxic potential), adefovir or probenecid. These agents must be discontinued at least 30 days prior to starting study medications. Brief course of aminoglycosides within 30 days of enrollment may be allowed after discussion with Study Chairs.
19. Concomitant Medications:

    * The following medications are expressly prohibited during the course of the trial: Astemizole, cisapride, ergot derivatives, hydroxyurea, midazolam, thalidomide, triazolam, vincristine, zalcitabine, ribavirin, doxorubicin, Voriconazole, St. John's wort or any medications that are contraindicated for concomitant use as described in the current product information packet insert for the ARV therapies used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2005-01; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Gay, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - The University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gay CL, Willis SJ, Cope AB, Kuruc JD, McGee KS, Sebastian J, Crooks AM, McKellar MS, Margolis DM, Fiscus SA, Hicks CB, Ferrari G, Eron JJ; Duke-UNC Acute HIV Infection Consortium. Fixed-dose combination emtricitabine/tenofovir/efavirenz initiated during acute HIV infection; 96-week efficacy and durability. AIDS. 2016 Nov 28;30(18):2815-2822. doi: 10.1097/QAD.0000000000001255. PMID 27662549
- [Result] Gay CL, Mayo AJ, Mfalila CK, Chu H, Barry AC, Kuruc JD, McGee KS, Kerkau M, Sebastian J, Fiscus SA, Margolis DM, Hicks CB, Ferrari G, Eron JJ; Duke-UNC Acute HIV Infection Consortium. Efficacy of NNRTI-based antiretroviral therapy initiated during acute HIV infection. AIDS. 2011 Apr 24;25(7):941-9. doi: 10.1097/QAD.0b013e3283463c07. PMID 21487250

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals with acute HIV (AHI) detected via a statewide AHI screening program in publicly funded sites and primary care sites are reported to the NC Department of Health and Human Services (DHHS). DHHS staff immediately refer acute cases to HIV care. From Jan 2005 and Dec 2011, all AHI cases referred to UNC and Duke were offered enrollment.
Pre-assignment Details: This was a single-arm, open-label study of emtricitabine/tenofovir/efavirenz started at enrollment. All participants received the same study treatment. Study treatment was not delayed for baseline resistance testing. Participants with transmitted baseline resistance to any drug in the regimen were followed on study on an alternative regimen.
Groups:
- Acute HIV Infection Treatment Group: This study was a dual-center, single-arm open-label study of the safety and efficacy of once daily, FTC/TDF/EFZ administered to participants with acute HIV infection
Period: Overall Study
Arm/Group | Acute HIV Infection Treatment Group
Started | 92
Completed | 90
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 92
Age, Categorical [Count of Participants; unit: Participants] — age (years) at time of acute HIV diagnosis
  Participants
    <=18 years | 0
    Between 18 and 65 years | 91
    >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] — Age at enrollment
  years | 27 [18 to 66]
Sex: Female, Male [Count of Participants; unit: Participants] — Gender at birth was determined at screening.
  Participants
    Female | 11
    Male | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 90
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 54
  White | 38
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — All participants were enrolled at either The University of North Carolina or Duke University.
  Participants
    United States | 92
CD4 cell count [Median (Full Range); unit: cells/mm^3] — Baseline CD4 cell count
  cells/mm^3 | 487 [13 to 1316]
HIV RNA level [Median (Full Range); unit: copies/mL] — baseline HIV RNA level
  copies/mL | 614898 [615 to 29807640]
Sexual risk group [Count of Participants; unit: Participants]
  Female | 11
  Heterosexual Male | 9
  Men who have sex with men | 72
sexually transmitted diseases within 8 weeks prior to diagnosis [Count of Participants; unit: Participants] — Diagnosis of sexually transmitted disease within the 8 weeks prior to diagnosis with acute HIV
  Participants | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Without Virologic Failure at Week 24
Description: Number of participants with a HIV RNA level <200 copies/mL at week 24
Time Frame: HIV RNA level prior to or at week 24 following enrollment
Measure: Count of Participants; unit: Participants
Groups:
- Acute HIV Infection Treatment Group: Participants suppressed to <200 copies/mL prior to or at week 24
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 90
Participants | 81

2. Secondary Outcome: Number of Participants Without Virologic Failure at Week 48
Description: HIV RNA level <50 copies/mL at week 48
Time Frame: HIV RNA level at week 48 following enrollment
Measure: Count of Participants; unit: Participants
Groups:
- Acute HIV Infection Treatment Group: Participants suppressed to <50 copies/mL prior at week 48
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 90
Participants | 71

3. Secondary Outcome: Number of Participants With HIV RNA Suppression at Week 96
Description: Number of participants wtih HIV RNA level <50 copies/mL at week 96
Time Frame: HIV RNA level at 96 weeks following enrollment
Measure: Count of Participants; unit: Participants
Groups:
- Acute HIV Infection Treatment Group: Participants who remained on study with viral suppression at week 96
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 75
Participants | 65

4. Secondary Outcome: Number of Participants With Baseline Genotypic Resistance to Antiretroviral Medications
Description: Prevalence of any of the surveillance drug resistance mutations associated with resistance to antiretroviral medications listed by the World Health Organization
Time Frame: At enrollment
Measure: Count of Participants; unit: Participants
Groups:
- Acute HIV Infection Treatment Group: Acute HIV infection treatment group
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 92
Participants | 17

5. Secondary Outcome: Number of Participants With Baseline Genotypic Resistance to One or More Antiretroviral Drugs in the Study Treatment
Description: Baseline genotypic resistance defined as presence of any surveillance drug resistance mutation to any drug in the study treatment listed by the World Health Organization
Time Frame: At enrollment
Measure: Count of Participants; unit: Participants
Groups:
- Acute HIV Infection Treatment Group: Baseline resistance testing was performed on all participants at enrollment.
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 90
Participants | 71

6. Secondary Outcome: Time to HIV RNA Suppression <50 Copies/mL
Description: Number of days from ART initiation to HIV RNA suppression <50 copies/mL
Time Frame: Number of days from start of study treatment until HIV RNA suppression, assessed through week 96
Measure: Median (Full Range); unit: days
Groups:
- Acute HIV Infection Treatment Group: Participants who remained on treatment at designated time points.
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 89
days | 105 [14 to 523]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant over the 96 weeks of the study.
Description: Adverse events were assessed at each visit and graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatrics Adverse Events.
Groups:
- Acute HIV Infection Treatment Group: Single-arml study of once daily emtricitabine/tenofovir/efavirenz administered to participants with acute HIV infection
Arm/Group | Acute HIV Infection Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 52/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acute HIV Infection Treatment Group (N=90)
Abdominal Discomfort (Gastrointestinal disorders) | 2 (2)
Abdominal Distension (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 3 (3)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1)
Abnormal Dreams (Psychiatric disorders) | 9 (11)
Alanine Aminotransferase Increased (Investigations) | 4 (4)
Anger (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (5)
Aspartate Aminotransferase Increased (Investigations) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Balance Disorder (Nervous system disorders) | 8 (8)
Blood Cholesterol Increased (Investigations) | 3 (4)
Blood Triglycerides Increased (Investigations) | 1 (1)
Claustrophobia (Psychiatric disorders) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2)
Depressed Mood (Psychiatric disorders) | 2 (3)
Depression (Psychiatric disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 7 (8)
Disturbance in Attention (Nervous system disorders) | 4 (4)
Dizziness (Nervous system disorders) | 25 (30)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Euphoric Mood (Psychiatric disorders) | 1 (1)
Eye Swelling (Eye disorders) | 1 (1)
fatigue (General disorders) | 4 (4)
Feeling Abnormal (General disorders) | 3 (3)
Feeling Drunk (General disorders) | 2 (2)
Feeling Jittery (General disorders) | 4 (4)
Flatulence (Gastrointestinal disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hangover (General disorders) | 1 (1)
Headache (Nervous system disorders) | 12 (15)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Initial Insomnia (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 12 (12)
Irritability (Psychiatric disorders) | 3 (3)
Lip Swelling (Gastrointestinal disorders) | 1 (1)
Lipase Increased (Infections and infestations) | 2 (2)
Low Density Lipoprotein Increased (Investigations) | 2 (2)
Memory Impairment (Nervous system disorders) | 1 (1)
Mood Swings (Psychiatric disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 16 (16)
Neutrophil Count Decreased (Investigations) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Obsessive Thoughts (Psychiatric disorders) | 1 (1)
Poor Quality Sleep (Nervous system disorders) | 1 (1)
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritis Generalised (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 6 (11)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 2 (6)
Rash Papular (Skin and subcutaneous tissue disorders) | 3 (3)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 (3)
Sleep Disorder (Psychiatric disorders) | 1 (1)
Sluggishness (General disorders) | 1 (1)
Somnolence (Nervous system disorders) | 9 (9)
Swelling Face (Skin and subcutaneous tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tunnel Vision (Nervous system disorders) | 1 (1)
Unevaluable Event (General disorders) | 3 (3)
Vision Blurred (Eye disorders) | 1 (1)
Visual Field Defect (Nervous system disorders) | 1 (1)
Visual Impairment (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes